CLINICAL TRIAL: NCT01089309
Title: Effect of Aldosterone Blockade on Metabolic Parameters and Arterial Compliance
Brief Title: Effect of Aldosterone Blockade on Arterial Compliance
Acronym: RAAS LAEI SAEI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WolfsonMC-2004-388
Record Dates: First submitted 2010-03-07; First posted 2010-03-18 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Arterial Stiffness; Arterial Elasticity
Keywords: Aldosterone Blockade; Arterial elasticity; Glycemic control
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aldosteron blokade, Arterial stiffness, Glucose homeostasis (Experimental)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — Spironolactone orally, at a dose of 50 mg/day for 12 months

SUMMARY:
The present study investigated the long-term (12 months) effect of spironolactone treatment on glucose homeostasis, metabolic parameters and vascular properties.

ELIGIBILITY:
Inclusion Criteria:

1. patients with type 2 diabetes mellitus

Exclusion Criteria:

1. history of unstable angina, myocardial infarction (MI), cerebrovascular accident (CVA)
2. major surgery within the six months preceding entrance to the study
3. unbalanced endocrine disease
4. any disease that might affect absorption of medications
5. plasma creatinine >2.5 mg/dl
6. elevation of liver enzymes to more that twice the upper normal limit
7. plasma potassium levels >5.5 mg/dl

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel